CLINICAL TRIAL: NCT05719012
Title: Efficacy and Safety of Umbilical Cord Mesenchymal Stem Cells in the Treatment of Long COVID-19: a Randomized, Double-blind, Parallel-controlled Study
Brief Title: Efficacy and Safety of Umbilical Cord Mesenchymal Stem Cells in the Treatment of Long COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in Recruitment
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DFSC-2023(CR)-02
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Long COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UC-MSCs (Experimental): UC-MSCs
  Interventions: Biological: UC-MSCs
- Placebo (Placebo Comparator): 0.9% Normal Saline
  Interventions: Biological: UC-MSCs

INTERVENTIONS:
Biological: UC-MSCs — Intravenous injection three times with one-month interval

SUMMARY:
To explore the efficacy and safety of Umbilical cord mesenchymal stem cells in the treatment of long COVID-19

ELIGIBILITY:
Inclusion Criteria:

1. The age ranges from 18 to 85 (inclusive), regardless of gender.
2. Patients with Confirmed SARS-CoV-2 infection, according to the consensus of the Chinese diagnostic criteria for COVID-19 (Tentative tenth Edition).
3. Patients with symptoms of long COVID-19 3 months from the onset of COVID-19, lasting for at least 2 months, and the symptoms cannot be explained by other diseases.
4. Be expected to live longer than 1 year.
5. Volunteer to participate in this clinical study and sign the written informed consent.

Exclusion Criteria:

1. Those who are using immunosuppressive drugs or long-term immunosuppressive drugs after organ transplantation.
2. T lymphocyte abnormality, HIV positive.
3. Highly allergic or have a history of severe allergy.
4. Pregnant and lactating women.
5. Patients with severe autoimmune disease history;
6. Patients with uncontrolled chronic diseases or serious complications;
7. Patients with malignant tumors;
8. Patients with pulmonary embolism, acute coronary syndrome, cerebral embolism or at high risk of thromboembolism;
9. Patients with severe organ dysfunction
10. Other situations that the researchers think are not suitable for participating in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Six min walking distances | Changes from baseline index at Day 30, Day 60, Day 90 and Day 180
  The maximum distance a person can walk in 6 min and acts as an endurance walking measure.
Lung function | Changes from the baseline index at Day 30, Day 60, Day 90 and Day 180
  The lung function assessed using FEV1, FEV1/FVC and DLco

SECONDARY OUTCOMES:
Changes of the levels of Inflammatory cytokines | Changes from the baseline levels at Day 30, Day 60, Day 90 and Day 180
  The levels of Inflammatory cytokines
Changes of the scores of Multidimensional Fatigue Inventory | Changes from the baseline scores at Day 30, Day 60, Day 90 and Day 180
  The degree of fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hosptial, Shanghai, China

IPD SHARING:
Plan to Share IPD: No